CLINICAL TRIAL: NCT06561178
Title: Individualized Tumor-Informed Circulating Tumor DNA (ctDNA) Analysis for Monitoring Postoperative Recurrence Following Neoadjuvant Therapy in Esophageal Squamous Cell Carcinoma (NEOCRTEC2401)
Brief Title: Individualized Tumor-Informed CtDNA Analysis for Monitoring Postoperative Recurrence in ESCC (NEOCRTEC2401)
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yang Hong, Prof., Sun Yat-sen University
Other Study IDs: B2024-302-01
Record Dates: First submitted 2024-08-12; First posted 2024-08-19 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: ctDNA; recurrence detection; esophageal squamous cell carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: molecular residual disease detection — ctDNA detection

SUMMARY:
The goal of this observational study or is to explore the correlation between dynamic changes in postoperative circulating tumor DNA (ctDNA) and recurrence risk using a novel, tumor-informed ctDNA detection technique, thus laying the foundation for further promoting ctDNA detection to guide postoperative adjuvant therapy decisions. This study focuses on patients with esophageal squamous cell carcinoma who did not achieve pCR following neoadjuvant therapy combined with surgical resection. The main question it aims to answer is:

Is there a correlation between postoperative ctDNA changes and tumor recurrence?

Participants will be asked to undergo postoperative ctDNA detection.

ELIGIBILITY:
Inclusion Criteria:

1. Operable locally advanced esophageal squamous cell carcinoma;
2. Have received neoadjuvant chemoradiotherapy ± immunotherapy and have not achieved pCR after R0 resection;
3. Can tolerate postoperative adjuvant immunotherapy;
4. Sufficient baseline tumor tissue and blood samples available for NGS testing;
5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1;
6. Consents to and is capable of complying with the scheduled study visits, treatment plans, laboratory tests, and other study procedures
7. Expected postoperative survival time of ≥ 6 months.

Exclusion Criteria:

1. Concurrent other malignant tumors;
2. Lack of a detailed histopathological diagnostic report for determining the nature of the lesion;
3. Severe and/or poorly controlled medical conditions that, in the investigator's judgment, could affect participation or interfere with study results;
4. Any social/psychological issues that, in the investigator's judgment, make the patient unsuitable for participation;
5. Unable to undergo long-term, regular postoperative follow-up at the current medical institution;
6. Unwilling or unable to comply with the study protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with esophageal squamous cell carcinoma who have not achieved pCR following neoadjuvant chemoradiotherapy and surgery.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between the recurrence of patients and the quantitative measurement of circulating tumor DNA (ctDNA) concentration. | 3 years
  Correlation were evaluated based on the sensitivity and specificity of ctDNA in predicting recurrence.The sensitivity and specificity were determined by evaluating the association between positive ctDNA and tumor recurrence.

SECONDARY OUTCOMES:
Postoperative molecular residual disease (MRD) positive rate | 3 years
Correlation between ctDNA detection and postoperative adjuvant therapy. | 3 years
  The ctDNA assay was employed to inform postoperative adjuvant therapy, with the objective of determining its potential to enhance patient prognosis.
correlation between patients' prognosis and landmark MRD status | 3 years
  The sensitivity and specificity were determined by evaluating the association between positive landmark MRD status and patients' prognosis.
2-year disease-free survival | 2 years
3-year disease-free survival | 3 years
5-year disease-free survival | 5 years
2-year overall survival | 2 years
3-year overall survival | 3 years
5-year overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Hong Yang, M.D.;Ph.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No